CLINICAL TRIAL: NCT06686485
Title: cOncomitant Left Atrial aPpendage Closure and Pulsed Field ablaTION-Asia
Acronym: OPTION-A
Status: Recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PF316
Record Dates: First submitted 2024-11-08; First posted 2024-11-13 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Concomitant Procedures; Atrial Fibrillation; PFA; LAAC
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment Subjects: A subject is considered enrolled once an approved informed consent form has been signed and dated. Enrolled Subjects will undergo AF ablation procedure with the FARAPULSE PFA System, followed by WATCHMAN implant during the same procedure.
  Interventions: Device: FARAPULSE™ PFA system and WATCHMAN LAAC Delivery Systems

INTERVENTIONS:
Device: FARAPULSE™ PFA system and WATCHMAN LAAC Delivery Systems — The FARAPULSE™ PFA System consists of the FARAWAVE™ Pulsed Field Ablation Catheter, the FARASTAR™ Pulsed Field Ablation Generator, and the FARADRIVE™ Steerable Sheath.
  The WATCHMAN LAA Closure Technology consists of the WATCHMAN Access System (which consists of the Access Sheath and Dilator and the WATCHMAN Delivery System (which consists of the delivery catheter and the pre-loaded closure device). The WATCHMAN Access System and WATCHMAN Delivery System permit device placement in the LAA via femoral venous access and crossing the inter-atrial septum into the left atrium.

SUMMARY:
Subjects enrolled in the OPTION-A study will be clinically indicated for atrial fibrillation (AF) ablation procedure with the FARAPULSE™ PFA system and treatment with WATCHMAN LAAC Device, per physician's medical judgement and according to hospitals' standard of care during the same procedure.

DETAILED DESCRIPTION:
The OPTION-A Study is an observational, prospective, single-arm, multi-center non-mandated post-market study. Subjects enrolled in the OPTION-A study will be clinically indicated for atrial fibrillation (AF) ablation procedure with the FARAPULSE PFA system and treatment with WATCHMAN LAAC Device, per physician's medical judgement and according to hospitals' standard of care. The objective(s) of the OPTION-A Study is to evaluate safety and effectiveness of catheter ablation with the FARAPULSE™ Pulsed Field Ablation (PFA) System and subsequent implant of Left Atrial Appendage closure (LAAC) with the WATCHMAN™ LAA Closure device in a concomitant procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically indicated for treatment with both the FARAPULSE™ PFA system and with WATCHMAN for LAAC, per physician medical judgement and as per hospitals' standard of care.
2. Subjects who are willing and able to provide informed consent.
3. Subjects who are willing and able to participate in all testing associated with this clinical study at an approved clinical investigational center.
4. Subjects whose age is 18 years or above, or who are of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

1. Subjects who underwent prior AF ablation procedure.
2. Subjects with atrial fibrillation that is secondary to electrolyte imbalance, thyroid disease, alcohol, or other reversible / non-cardiac causes.
3. Already surgically closed or otherwise excluded LAA.
4. The LAA anatomy does not accommodate a Closure Device.
5. Known or suspected atrial myxoma.
6. Presence of intracardiac thrombus.
7. Subjects with a current interatrial baffle or patch, history of atrial septal repair or has an ASD/PFO device.
8. Subjects with a presence of a mechanical valve prosthesis in any position.
9. Subjects with a myocardial infarction within 30 days prior to enrollment.
10. Subjects had a prior stroke (of any cause, whether ischemic or hemorrhagic) or transient ischemic attack (TIA) within the 90 days prior to enrollment.
11. Any planned electrical cardioversion within 30 days following LAAC device implant.
12. Subjects with a known inability to obtain vascular access.
13. Subjects with any contraindication to percutaneous catheterization procedure (e.g., patient size does not accommodate required catheters, ventriculotomy or atriotomy), active conditions (e.g. infection, bleeding disorder, unstable angina) or congenital abnormalities (severe rotational anomalies of the heart or great vessels) are present*.
14. Subjects with any contraindications to short term use of anticoagulation therapy, or aspirin for conditions different from atrial fibrillation.
15. Subjects who are pregnant or planning to be pregnant.
16. Subjects with a life expectancy of ≤ 1 year per investigator's opinion.
17. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments. Each instance must be reviewed by the sponsor to determine eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects enrolled in the OPTION-A study will be clinically indicated for an Atrial Fibrillation ablation procedure utilizing the FARAPULSE PFA System as well as implantation of the WATCHMAN device per physician's medical judgement, and according to the hospitals' standard of care during the same procedure. The subjects selected for participation in the study will be from the investigator's general patient population. The investigator or designee has the responsibility for screening all potential subjects and selecting those who meet study eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 433 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Periprocedural or procedure-related Composite Serious Adverse Events will be assessed | 30 days post index procedure
  The primary safety endpoint (PSE) is the proportion of subjects with one or more of the periprocedural device or procedure-related Composite Serious Adverse Events (CSAEs) assessed at 30 days following the Index Procedure.
Acute Treatment Success will be assessed | between index procedure and 30 days post index procedure
  The primary effectiveness endpoint (PEE) is the proportion of subjects with Acute Treatment Success assessed among those receiving ≥1 PFA application and who have a WATCHMAN attempted or implanted.

SECONDARY OUTCOMES:
Device or procedure-related Composite Serious Adverse Events (CSAEs) assessed | 1 year post index procedure
  Device or procedure-related Composite Serious Adverse Events (CSAEs) assessed at 360 days following the Index Procedure

CONTACTS AND LOCATIONS:
Locations (27):
- China (8):
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Beijing Anzhen Hospital of the Capital University of Medical Sciences, Beijing
  - Huaxi Hospital of Sichuan University, Chengdu
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou
  - QiLu Hospital of ShanDong University, Jinan
  - Shanxi Cardiovascular Hospital, Taiyuan
  - Zigong First People's Hospital, Zigong
- Hong Kong (4):
  - Prince of Wales Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Queen Elizabeth Hospital, Kowloon
- Japan (9):
  - Shonan Kamakura General Hospital, Kamakura-shi, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Kurashiki Central Hospital, Kurashiki-shi, Okayama Kurashiki-shi
  - Saitama Red Cross Hospital, Saitama, Saitama
  - Sakakibara Heart Institute, Sakakibara Heart Foundation, Fuchu-shi, Tokyo
  - Kokura Memorial Hospital, Fukuoka-ken
  - Yokosuka Kyosai Hospital, Kanagawa
  - Toho University Ohashi Medical Center, Meguro-ku
  - Osaka Keisatsu Hospital, Osaka
- Malaysia (2):
  - Institute Jantung Negara, Kuala Lumpur
  - Pusat Jantung Sarawak, Kuching
- Asian Heart and Vascular Centre, Singapore, Singapore
- Taiwan (3):
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No